CLINICAL TRIAL: NCT02297256
Title: Prospective Study of Thoracolumbar Spinal Fusion Graft Efficacy: Bone Marrow Aspirate Concentrate Versus Iliac Crest Bone Graft
Brief Title: Prospective Study of Thoracolumbar Spinal Fusion Graft
Acronym: BMAC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12-02411
Record Dates: First submitted 2014-10-02; First posted 2014-11-21 (Estimated); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Lumbar Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Transplantation, Homologous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BMAC & Allograft (Active Comparator): Subjects will be treated with bone marrow aspirate concentrate (BMAC) and allograft during posterior lumbar/lumbosacral spinal fusion. During lumbar spine surgery, 12 teaspoons of bone marrow will be taken (aspirated) from one side of hip bone. This may be repeated on the other side of hip bone for a total of 12, 24, or 36 teaspoons of bone marrow total taken from your hip bone depending on the decision made by the surgeon. The bone marrow will then be concentrated with a machine for 15 minutes to a final volume of 2, 4, or 6 teaspoons of BMAC. BMAC will be combined with packed allograft bone chips using another machine to produce two or three constructed bone logs. The bone logs will be laid along the backside of the spine and between each vertebral body.
  Interventions: Procedure: BMAC & Allograft
- Iliac Crest Bone Graft (Active Comparator): Subjects who are in the Iliac Crest Bone Graft arm will be treated with Iliac crest bone grafts (ICBG) during posterior lumbar/lumbosacral spinal fusion. During lumbar spine surgery, the surgeon will make an incision to expose the iliac crest (hip bone), and cutting out the segments of the bone that will be needed, based on the decision of the surgeon. The bone chips will be laid along the backside of the spine and also between each vertebral body where the bone will fuse into place. When the bone becomes solid/fused, there is no movement in the fused spine.
  Interventions: Procedure: Iliac Crest Bone Graft

INTERVENTIONS:
Procedure: BMAC & Allograft — Use of Allograft infused with adult stem cells from the bone marrow aspirate harvested from the iliac crest during posterior lumbar/lumbosacral spinal fusion.
  Other Names: Bone Marrow Aspirate Concentrate & Allograft
  Arms: BMAC & Allograft
Procedure: Iliac Crest Bone Graft — Use of iliac crest bone grafts (ICBG) during posterior lumbar/lumbosacral spinal fusion.
  Other Names: ICBG
  Arms: Iliac Crest Bone Graft

SUMMARY:
This study is a single-center, prospective randomized clinical study intended to compare and evaluate the efficacy of subjects who are treated with bone marrow aspirate concentrate (BMAC) and allograft to iliac crest bone grafts (ICBG) during posterior lumbar/lumbosacral spinal fusion.

DETAILED DESCRIPTION:
Subjects who are candidates for posterior lumbar or lumbosacral spinal fusion without anterior interbody support will be screened for inclusion in the study. Participants will be enrolled and randomized to either the BMAC + allograft or ICBG group. An enrollment ratio of two BMAC + allograft to one ICBG subject (2:1) for up to a total of 40 subjects will be enrolled in the study which also accounts for failed screening subjects. The study will determine and compare differences in fusion rate and health related quality of life parameters at 6 weeks, 3 months, 6 months, 1 year, and 2 years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years old or older
* Scheduled for elective posterior spinal fusion of the thoracolumbar spine or lumbar spine with or without anterior interbody support
* Failed at least 6 weeks of conservative care
* ODI v2.1 score > 30%
* No contraindication to BMAC (as per manufacturer)
* Signed consent form

Exclusion Criteria:

* Spondylolisthesis grade ≥ 3
* Pagets disease, osteomalacia, or any metabolic bone disease
* Use of medications that interfere with bone healing (chronic steroids)
* Patient unlikely to comply with post-op schedule with physician
* Recent history of chemical dependency
* Participation in other investigational device trial(s) within past 30 days
* Active malignancy
* Pregnancy or planning to become pregnant
* Direct involvement in execution of this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
CT scan to assess fusion status | Pre-operative, Post Operative 1 Year
Oswestry Disability Index (ODI) | Pre-operative, Post Operative 1 Year
Short Form Health Survey (SF-12) | Pre-op, Post Operative 1 Year
Numeric Pain Rating Scale | Pre-op, Post Operative 1 Year
Length of Stay | Post Operative 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Passias, MD, Principal Investigator — NYU School of Medicine
Locations (3):
- United States (3):
  - NYU Hospital for Joint Diseases, New York, New York
  - Center for Musculoskeletal Care (CMC), New York, New York
  - NY Spine Institute, Westbury, New York

REFERENCES:
- [Background] Asahara T, Masuda H, Takahashi T, Kalka C, Pastore C, Silver M, Kearne M, Magner M, Isner JM. Bone marrow origin of endothelial progenitor cells responsible for postnatal vasculogenesis in physiological and pathological neovascularization. Circ Res. 1999 Aug 6;85(3):221-8. doi: 10.1161/01.res.85.3.221. PMID 10436164
- [Background] Gan Y, Dai K, Zhang P, Tang T, Zhu Z, Lu J. The clinical use of enriched bone marrow stem cells combined with porous beta-tricalcium phosphate in posterior spinal fusion. Biomaterials. 2008 Oct;29(29):3973-82. doi: 10.1016/j.biomaterials.2008.06.026. Epub 2008 Jul 18. PMID 18639333